CLINICAL TRIAL: NCT05210504
Title: Determinants of Alpha-aminoadipic Acid (2-AAA) and Relationship to Diabetes: Study 3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jane Ferguson, Associate Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Lysine study #3
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: lysine
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Lysine; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants administered oral lysine (Experimental): participants will be administered 5g oral lysine
  Interventions: Drug: L-Lysine; Drug: Normal Saline

INTERVENTIONS:
Drug: L-Lysine — 5g L-lysine in 50ml water, administered orally
Drug: Normal Saline — Normal (0.9%) Saline

SUMMARY:
This study aims to assess the effect and breakdown of lysine administration, specifically examining whether it leads to increased plasma 2-AAA in healthy humans.

DETAILED DESCRIPTION:
The purpose of this study is to investigate a novel biomarker, α-aminoadipic acid (2-AAA), which may influence the risk of diabetes. 2-AAA has been identified as a novel predictor of diabetes development in humans, identifying at-risk individuals before any detectable glucose abnormalities. 2-AAA is a naturally occurring metabolite in the body, and it has no known adverse effects at normal physiological levels. 2-AAA is generated in the body from the breakdown of lysine. Lysine is one of the twenty essential amino acids, meaning that it is essential for human function, but that our body cannot manufacture it. Thus, it is acquired from dietary sources (such as meat, eggs, soybeans and legumes), with a recommended daily intake of 30 mg/kg/day. Amino acids are the building blocks of proteins, which are what allow our cells, organs and body to maintain structure and function. The investigators are interested in whether 2-AAA is increased in the body after consumption of lysine.

ELIGIBILITY:
Inclusion Criteria:

-Prior participant in 2-AAA Dietary study.

Exclusion Criteria:

* Newly diagnosed disease, including cardiovascular, renal, liver disease, or Diabetes mellitus.
* Individuals who are pregnant or lactating.
* Inability to provide written or electronic informed consent.
* Inability to fast for 8 hours.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Ferguson, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We enrolled 23 individuals to the study. 4 individuals withdrew before the start of the study due to scheduling conflicts, and 2 individuals were lost to follow up.
Period: Overall Study
Arm/Group | Participants Administered Oral Lysine
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All individuals are analyzed where possible. One participant did not provide a baseline blood draw, and was excluded from the analysis for plasma measurements.
Arm/Group | Participants Administered Oral Lysine
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Level of 13C 2-AAA in Plasma
Description: Alpha aminoadipic acid (2-AAA) concentration determined through mass spectrometry, quantified to standard. The change was calculated as the area under the curve from baseline to 6 hours post-lysine administration of isotope labeled 2-AAA.
Time Frame: Baseline to 6 Hours post-lysine administration
Population: One individual missed their baseline and 1Hr blood draws, and was omitted from the analysis.
Measure: Mean (Standard Deviation); unit: uM*Hr
Arm/Group | Participants Administered Oral Lysine
Number analyzed (Participants) | 16
uM*Hr | 1.742 (0.611)

2. Primary Outcome: Change in Level of 2-AAA in Urine
Description: Alpha aminoadipic acid (2-AAA) concentration determined through mass spectrometry, quantified to standard. The change was calculated as the total amount of 13C 2-AAA in micromoles excreted from Baseline to 6 hours.
Time Frame: Baseline to 6 Hours post-lysine administration
Population: For one individual the volume of urine was not recorded, and their data could not be analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles
Arm/Group | Participants Administered Oral Lysine
Number analyzed (Participants) | 16
Micromoles | 7.69 (4.25)

ADVERSE EVENTS:
Time Frame: Data were collected throughout the 6 hour study period.
Arm/Group | Participants Administered Oral Lysine
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT05210504/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/04/NCT05210504/ICF_000.pdf